CLINICAL TRIAL: NCT04402671
Title: Lateral Ridge Augmentation Using Cross-linked or Non-cross-linked Collagen Membrane: a Pilot Randomized Clinical Trial
Brief Title: Lateral Ridge Augmentation Using Cross-linked or Non-cross-linked Collagen Membrane
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saint-Joseph University (Other)
Responsible Party: Principal Investigator, Mario Haddad, Principal Investigator, Saint-Joseph University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMD188
Record Dates: First submitted 2020-05-15; First posted 2020-05-27 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Bone Loss
Keywords: Guided bone regeneration; collagen membrane; crosslinked collagen membrane; Bone augmentation
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Intervention Model Description: This study is a pilot randomized clinical trial with parallel groups, with an observation period of 6 - 9 months. It is set to identify the equivalence between the test and the control procedures. An equal randomization is set for the 2 groups
Who Masked: Participant, Outcomes Assessor
Masking Description: The patients are blind to the allocation. The radiographic volumetric changes and the histomorphometrical analysis are assessed by blind examiners.
  Random allocation was done by the sequentially sealed envelope method. At the time of membrane placement during the surgery, the envelope corresponding to the case sequence number is opened specifying the group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- non-crosslinked collagen membrane group (Active Comparator): 2 patients (1 male, 1 female)
  Interventions: Other: non-cross-linked porcine skin collagen membrane
- glutaraldehyde cross-linked collagen membrane (Active Comparator): 2 patients (2 females)
  Interventions: Other: glutaraldehyde cross-linked bovine collagen membrane

INTERVENTIONS:
Other: non-cross-linked porcine skin collagen membrane — non-cross-linked porcine skin collagen membrane used is Bioguide, Geistlisch Pharma AG, Wolhusen, Switzerland.
  Other Names: Bioguide
  Arms: non-crosslinked collagen membrane group
Other: glutaraldehyde cross-linked bovine collagen membrane — glutaraldehyde cross-linked bovine collagen membrane GCLM used is RTM Collagen®, Osteogenics Biomedical, Lubbock, TX, USA.
  Other Names: Cytoplast RTM
  Arms: glutaraldehyde cross-linked collagen membrane

SUMMARY:
The objective of the present trial is to test clinically, radiographically and histologically , in a lateral alveolar ridge augmentation model (without simultaneous implant placement) the efficiency in supporting bone formation of a glutaraldehyde cross-linked collagen membrane compared to a non-cross-linked collagen membrane with the use of a composite autograft-xenograft mix prepared in a 1:3 ratio

DETAILED DESCRIPTION:
This study is a pilot one, no sample size calculation has been performed. Random allocation was done by the sequentially sealed envelope method.

Interventions

Pre-operative preparation:

* Scaling and root planning and delivering proper hygiene instructions.
* Fabrication of the occlusal stent/radiographic guide (Silicone impression of the concerned arch and pouring of the model. Denture teeth are added on the edentulous space of the cast. A 2 mm thickness clear resin sheet is adapted to the cast with a vacuum forming machine. The borders of the stent are trimmed with a tungsten carbide bur to remove the parts that are covering the soft tissues. At the level of the surgical site, the intaglio of the guide is reduced in a way to prevent any interference with the swollen soft tissues during the one-week CBCT assessment. In the middle of each denture tooth, 2 mm cylindrical holes are created occlusally. Gutta-percha is inserted in these holes to serve as radio-opaque markers and as reference points for per-operative measurements.
* Pre-operative Cone Beam CT (CBCTpreop) with the radiographic guide/occlusal stent in the mouth

Surgical intervention:

Patients are put on an antibiotic regimen consisting of 1 g co-amoxiclav taken twice daily (Augmentin, GlaxoSmithKline, Brentford, United Kingdom), starting the evening prior to surgery and continued for 10 days. For patients allergic to penicillins, Clindamycin 300 mg taken every 6 hours (Dalacin C, Pfeizer, New York City, NY, USA) is prescribed. Before surgery, the patient is asked to rinse with 0.12% chlorhexidine solution for one minute. Local anesthesia is delivered using 4% articaine with epinephrine 1:100,000 (Septanest, Septodont, Saint Maur des Fosses, France). After mid-crestal and vertical releasing incisions are being made, full thickness flaps are raised. The recipient bone is curetted to remove any soft tissue that may impede bone healing. Using a ridge mapping caliper, Crestal Bone Width is recorded at 1 (CBWpreop1), 3 (CBWpreop3) and 5 (CBWpreop5) mm from the crest at the level of the gutta-percha markers of the guide. Using a periodontal probe, another measure is recorded from the Ridge Crest to the Border of the Guide (RC-BG). This measure will be used at the 6-month re-entry to locate the vertical position of the pre-operative ridge mapping measurements in case of vertical bone changes. On the buccal flaps, superficial periosteal releasing incisions are performed to release the flap tension and to access the submucosal tissues. Once accessed, the submucosal tissues are stretched by inserting the wide end of a periosteal elevator into the incision line and pushing it in a coronal direction, resulting in flap elongation. In the posterior mandible, the lingual flap is elongated by a lateral stretching movement using the wide end of the periosteal elevator to separate the sub-mucosal tissues from the underlying muscle. More anteriorly in the mandible, a superficial periosteal incision is performed in the lingual flap. The buccal aspect of the crest is decorticated to ensure vascularization at the recipient site. The particulate bone graft consisting of a composite autograft-xenograft is then prepared in a 1:3 ratio mixed in sterile saline. A 0.5 cc spoon is used to have an exact 1:3 ratio. The spoon is slightly overfilled, and the excess is eliminated with a spatula. Only the full spoon content is used in the bone graft mix. The autograft is obtained by scraping the adjacent bony region with a bone scraper (SafeScraper TWIST, META, Reggio Emilia, Italy). The xenograft used is an anorganic bovine bone mineral with a 250-1000 microns particle size (OCS-B Xenomatrix®, Nibec, Chungcheongbuk-do, Korea, available also under the name of Straumann Xenograft® and Creos Xenogain®). After opening the sequentially sealed envelope, the patient is allocated to test or control groups. In the test group a glutaraldehyde cross-linked bovine collagen membrane GCLM is used (RTM Collagen®, Osteogenics Biomedical, Lubbock, TX, USA), in the control group a non-cross-linked porcine skin collagen membrane is used (Bioguide, Geistlisch Pharma AG, Wolhusen, Switzerland). The membrane is fixed first on the buccal side with titanium pins (Masetrpin®, Meisinger, Neuss, Germany) in a way to create a pouch like space. Second, the composite graft is applied between the membrane and the crest with a slight over fill. Then the membrane is slightly stretched, wrapped over the ridge and tightly stabilized palatally/lingually with titanium pins. The graft-membrane complex should be completely immobile at finger pressure. A tight wound closure is achieved by placing a first line of horizontal mattress sutures followed by a second line of interrupted sutures along the horizontal incision. The vertical releasing incisions are closed with a combination of Laurel-Gottlow sutures and interrupted sutures. The sutures used are 4(0) PTFE monofilament sutures (Osteogenics Biomedical, Lubbock, TX, USA). Beside the antibiotic regimen described earlier, all patients are prescribed 0.12% chlorhexidine mouthwash (twice daily for 2 weeks, starting from the day after surgery), NSAIDs drugs (Bruffen 400mg every 6 hours, Abbott Laboratories, Illinois, CHI, USA) and/or paracetamol-opioid analgesics (Solpadeine, Omega Pharma Nazareth, Belgium). An extraoral cold pressure dressing is applied to minimize postoperative swelling. Sutures are removed 3 weeks after surgery.

During the first week after surgery, a Cone Beam CT (CBCTpostop) of the operated region is performed, with the radiographic guide in place.

Follow-up visits will be performed after 1, 3, 6, 10, 14, 18, 22 and 26 weeks.

Re-entry:

At 6 months post-surgery, another Cone Beam CT (CBCTre), with the same radiographic guide in place, is taken for bone volume assessment and for implant planning. Mid-crestal and vertical releasing incisions are made. Full thickness flaps are raised, and the pins are removed. Any non-integrated bone graft material is gently scraped and washed out with saline. The guide is put in place and using the previously recorded RC-BG measurement to correctly locate the level of the ridge crest before the ridge augmentation surgery, Crestal Bone Width is recorded with the ridge mapping caliper at the same locations (CBWre1, CBWre3, CBWre5) taken during the regeneration surgery. In addition, a UNC-15 periodontal probe is pushed with pressure against the ridge at a 45 degrees angle at the level of each gutta-percha marker and at 3 mm form the ridge top. The amount probe penetration in the grafted bone volume is recorded.

A 2 mm diameter trephine bone biopsy is collected for histomorphometrical and immunohistochemichal analysis. When possible, the biopsy is extracted horizontally from the buccal aspect of the ridge at 4 mm from the crest, otherwise it will be collected vertically from the ridge top. One biopsy is collected per patient, taken where the lateral ridge defect is the most severe.

Then the implants are inserted, at the prosthetically planned positions, according to the manufacturer's instructions. Flaps are sutured and a post-operative medication is prescribed consisting of an antibiotic coverage, an analgesic, and a chlorhexidine mouthwash.

Three months later, the implants are uncovered for abutment connection and will be subsequently restored.

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients, non-smokers or smokers<10 cigarettes/day.
* Age between 20 and 75.
* Full mouth bleeding score (FmBS) <20 %.
* Full mouth plaque score (FmPS) <15%.
* Presence of a residual alveolar ridge with residual bone width < 5 mm and adequate
* bone height in the maxilla and the mandible.
* Tooth extraction performed at least 6 weeks before surgery.
* Presence of enough teeth to support an occlusal stent/radiographic guide.

Exclusion Criteria:

* Systematic diseases.
* History of radiotherapy in the head and neck region in the last 5 years.
* Active periodontitis on the remaining teeth.
* Pregnancy.
* Allergy to collagen.
* Intake of medications that may have an effect on bone turnover and mucosal healing (i.e., tetracycline within the last month, steroids within the last 6 months, bisphosphonates or fluorides at bone therapeutic levels, vitamin D and metabolites at therapeutic levels within the last 6 months).

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Linear measurements outcomes | 6 - 9 months
  the ridge mapping changes in linear measurements between initial ridge width and reentry ridge width at 1, 3 and 5 mm from the ridge crest

SECONDARY OUTCOMES:
Volumetric measurements outcome | 6 - 9 months
  Pre-operative Cone Beam CT (CBCTpreop), a Cone Beam CT the first week after surgery (CBCTpostop), and a Cone Beam CT at re-entry post-surgery (CBCTre), with the radiographic guide/occlusal stent in the mouth, are taken.
  DICOM files from the 3 CBCT scans are uploaded to the BlueSky Plan software (BlueSkyBio, Grayslake, IL, USA) and are superimposed using the gutta-percha markers of the radiographic guide. The Region Of Interest (ROI) is delineated Vpreop, Vpostop and Vre are the volume in cubic millimeters of the ROI measured from the CBCTpreop, CBCTpostop and the CBCTre, respectively.
  The volumetric outcomes from the DICOM data are used for each group to calculate:
  * the volume of graft resorption.
  * the graft volume created after GBR
  * the bone volume gain.
the percentage of graft volume resorption. | 6 - 9 months
  The percentage of graft volume resorption is calculated by deviding the volume of the graft resorbtion on the volume created after GBR
Linear measurements outcomes on DICOM data | 6 - 9 months
  On each gutta percha site on the DICOM files these measurements are assessed:
  Linear measurements in millimeters at 1, 3, 5 mm from the ridge crest in a plane orthogonally bisecting the dental arch at the level of each gutta-percha marker, taken form the ROI of CBCTpreop and CBCTre respectively.
  The changes of the linear measurements outcomes on DICOM data between CBCTpreop and CBCTre.
Soft tissue healing | 6 - 9 months
  Soft tissue healing will be assessed during the follow-up visits for the following occurrences Redness and swelling. Wound dehiscence and membrane exposure. Infections or any other unaccounted complications will be recorded
Periodontal Probe Penetration (PP) | 6 - 9 months
  PP reflecting the amount of graft maturation is recorded and compared between sites and between patients.
Histology | 6 - 9 months
  Histology analysis of the bone biopsies taken from the regenerated crests at re-entry surgery
Histomorphometry: percentage of new bone formation | 6 - 9 months
  Calculation of Percentage new bone formation in the bone biopsies taken from the regenerated crests at re-entry
Histomorphometry: percentage of remaining graft particles | 6 - 9 months
  Calculation of the percentage remaining graft particles in the bone biopsies taken from the regenerated crests at re-entry
Histomorphometry: percentage of connective tissue | 6 - 9 months
  Calculation of the percentage of connective tissue in the bone biopsies taken from the regenerated crests at re-entry

CONTACTS AND LOCATIONS:
Overall Officials: Carole F Chakar, PhD, Study Director — Saint-Joseph University
Locations (1):
- Mario Haddad, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: As soon as the study is published
Access Criteria: A scientific journal